CLINICAL TRIAL: NCT01974947
Title: Relationship Between Sperm Parameters and Metabolic Syndrome in a Infertile Couple Partner Man
Brief Title: Metabolic Syndrome and Male Infertility
Acronym: Metasperme
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI 10033
Record Dates: First submitted 2013-07-26; First posted 2013-11-04 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Male Infertility
Keywords: Metabolic syndrome; Epigenetic; Male infertility; Sperm parameters; Biomarkers
MeSH Terms: conditions — Infertility, Male; Metabolic Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and sperm samples will be collected from all patients BLOOD :Whole blood was collected on dry, heparin or EDTA tubes. After several soft turnings, tubes were centrifuged at 1900g for 10min.Then plasma, serum, buffy coat or red blood cells were taken in microtubes and frozen at -80°C.
  SPERM: After liquefaction, total sperm was centrifuged at 600g for 10min. Seminal plasma was collected directly on microtubes and stored at -80°C. After trypsinisation, spermatozoa were fixed in Carnoy solution and stored at -20°C.
  DNA was separated from buffy coat using DNA extract kit
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infertile men: Man partner of an infertile couple. Blood sample, sperm sample and clinical examens will be done at the day of the inclusion
  Interventions: Other: Blood sample, sperm sample and clinical examens

INTERVENTIONS:
Other: Blood sample, sperm sample and clinical examens — Blood sample, sperm sample and clinical examens will be done at the day of the inclusion

SUMMARY:
Multidisciplinary, multicentric, cross-sectional study on men in infertile couples who conduct their sperm test through their diagnosis of infertility

DETAILED DESCRIPTION:
Assessment of sperm parameters and metabolic syndrome relations in men attending a Reproductive Biomedicine centre for an infertility of their couple.

Secondary objectives are to study relationship between sperm parameters and:

* adiposity and insulin resistance
* inflammation
* oxydative stress in blood and semen
* hormonal status Innovative parameters will also be assessed to determine the quality of semen (length of fingers, wrist circumference and epigenetics studies)

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years-old man
* man consulting for primary or secondary infertility, with or without earlier notion of paternity
* patient insured with a social security scheme
* patient who have had a prior medical consultation
* patient who have done informed and written consent to participate in the research study

Exclusion Criteria:

* patient with problems understanding French
* patient smoking more than two-pack-a-day
* patient monitoring for viral risk.
* man with an unidiopathic infertility which may be explained by:

  1) identifiable factors in direct questioning at the sperm analysis:
* exposure to toxic products
* infectious disease history
* pathological anatomical background 2) factors identified at the etiologic investigation: cytogenetic and genetic

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Man consulting for primary or secondary infertility, with or without earlier notion of paternity
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2013-07-18 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2016-01-20 (Actual)

PRIMARY OUTCOMES:
Number of spermatozoid and their relation with syndrome metabolic parameters | Day 0
  We will measure the parameters of metabolic syndrome (triglycerides, HDL and LDL cholesterol, systolic and diastolic blood pressure, fasting glucose) and correlate them with the number of spermatozoid .

SECONDARY OUTCOMES:
Relationship between spermogram and spermocytogram and other metabolic parameters | Day 0
  Relationship between other spermogram/spermocytogram and metabolic markers (biomarkers and anthropometric adiposity and insulin resistance)
Environmental parameters | Day 0
  Evaluation of environmental parameters (physical activity, tobacco consumption, quality of life) by classical questionnaire
Relationship between spermogram and spermocytogram and other metabolic parameters | Day 0
  Relationship between other spermogram/spermocytogram and markers of inflammation
Relationship between spermogram and spermocytogram and other metabolic parameters | Day 0
  Relationship between other spermogram/spermocytogram and markers of oxidative stress (plasma, seminal genetic polymorphisms involved in oxidative stress, genetic analyzes of sperm)
Relationship between spermogram and spermocytogram and other metabolic parameters | Day 0
  Relationship between other spermogram/spermocytogram and hormonal markers
Relationship between spermogram and spermocytogram and other metabolic parameters | Day 0
  Relationship between other spermogram/spermocytogram and innovative settings (studies epigenetic finger length and width of the wrist)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Lévy, MD, PhD, Principal Investigator — Tenon Hospital
Locations (1):
- Jean Verdier Hospital, Bondy, France

REFERENCES:
- [Background] Sermondade N, Faure C, Fezeu L, Shayeb AG, Bonde JP, Jensen TK, Van Wely M, Cao J, Martini AC, Eskandar M, Chavarro JE, Koloszar S, Twigt JM, Ramlau-Hansen CH, Borges E Jr, Lotti F, Steegers-Theunissen RP, Zorn B, Polotsky AJ, La Vignera S, Eskenazi B, Tremellen K, Magnusdottir EV, Fejes I, Hercberg S, Levy R, Czernichow S. BMI in relation to sperm count: an updated systematic review and collaborative meta-analysis. Hum Reprod Update. 2013 May-Jun;19(3):221-31. doi: 10.1093/humupd/dms050. Epub 2012 Dec 12. PMID 23242914
- [Background] Hammoud AO, Gibson M, Peterson CM, Meikle AW, Carrell DT. Impact of male obesity on infertility: a critical review of the current literature. Fertil Steril. 2008 Oct;90(4):897-904. doi: 10.1016/j.fertnstert.2008.08.026. PMID 18929048
- [Background] Sermondade N, Faure C, Fezeu L, Levy R, Czernichow S; Obesity-Fertility Collaborative Group. Obesity and increased risk for oligozoospermia and azoospermia. Arch Intern Med. 2012 Mar 12;172(5):440-442. doi: 10.1001/archinternmed.2011.1382. PMID 22412113
- [Background] Michalakis K, Mintziori G, Kaprara A, Tarlatzis BC, Goulis DG. The complex interaction between obesity, metabolic syndrome and reproductive axis: a narrative review. Metabolism. 2013 Apr;62(4):457-78. doi: 10.1016/j.metabol.2012.08.012. Epub 2012 Sep 20. PMID 22999785
- [Result] Bongrani A, Elfassy Y, Brun JS, Rame C, Mellouk N, Fellahi S, Bastard JP, Levy R, Vasseur C, Froment P, Dupont J. Expression of adipokines in seminal fluid of men of normal weight. Asian J Androl. 2019 Sep-Oct;21(5):528-530. doi: 10.4103/aja.aja_25_19. No abstract available. PMID 31115360
- [Result] Elfassy Y, Bongrani A, Levy P, Foissac F, Fellahi S, Faure C, McAvoy C, Capeau J, Dupont J, Feve B, Levy R, Bastard JP; Metasperme group. Relationships between metabolic status, seminal adipokines, and reproductive functions in men from infertile couples. Eur J Endocrinol. 2020 Jan;182(1):67-77. doi: 10.1530/EJE-19-0615. PMID 31705791
- [Derived] Saget S, Kappeler L, Grandjean V, Leneuve P, Berthaut I, Faure C, Czernichow S, Racine C, Levy R, Dupont C; Metasperme Collaboratif group. Association between metabolic disorders and seminal plasma miRNA levels: a pilot study. Basic Clin Androl. 2022 Jun 7;32(1):9. doi: 10.1186/s12610-022-00159-7. PMID 35668388